CLINICAL TRIAL: NCT00937495
Title: A Phase II Study of Suberoylanilide Hydroxamic Acid and Bortezomib in Advanced Soft Tissue Sarcomas
Brief Title: Vorinostat and Bortezomib in Treating Patients With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03810; MC0778; CDR0000646715; MAYO-MC0778; N01CM62205 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2013-09

CONDITIONS: Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Vorinostat; Bortezomib

ARMS (1):
- Treatment (vorinostat, bortezomib) (Experimental): Patients receive 400 mg vorinostat orally once daily on days 1-14. Patients also receive 1.3 mg/m^2 bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: bortezomib

INTERVENTIONS:
Drug: vorinostat — 400 mg given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: bortezomib — 1.3 mg/m^2 given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase II trial is studying how well giving vorinostat together with bortezomib works in treating patients with advanced soft tissue sarcoma. Vorinostat and bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vorinostat together with bortezomib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate in patients with advanced soft tissue sarcoma treated with vorinostat and bortezomib.

SECONDARY OBJECTIVES:

I. Characterize the toxicity of this regimen in these patients. II. Evaluate the progression-free survival and median overall survival of patients treated with this regimen.

OUTLINE:

Patients receive vorinostat orally (PO) once daily on days 1-14. Patients also receive bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 6 months for up to 2 years. (As of Addendum 7, patient follow-up no longer required.)

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced, unresectable, or metastatic soft tissue sarcoma (STS)
* Measurable disease, defined as >= 1 lesion that can be accurately measured in >= 1 dimension as >= 2 cm by conventional techniques OR >= 1 cm by spiral computed tomography (CT) scan
* No small round cell tumors, including the following:

  * Primitive neuroectodermal tumor
  * Rhabdomyosarcoma
  * Ewing sarcoma
  * Osteosarcoma
* No known active and/or untreated brain metastases and/or brain metastases requiring ongoing therapy (e.g., corticosteroids)

  * Treated, inactive brain metastases not requiring ongoing therapy allowed provided the brain metastases have been stable for >= 1 month as assessed by intracranial imaging AND there is no indication of increased vascularity of the treated metastases within 14 days before study entry as assessed by magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy >= 12 weeks
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin normal
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to take oral medication
* No peripheral neuropathy >= grade 2
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia or myocardial infarction within the past 6 months
  * Psychiatric illness and/or social situation that would limit compliance with study requirements
* No history of Torsades de Pointes
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to vorinostat or bortezomib
* No more than 1 prior systemic treatment for advanced STS, including investigational agents

  * Adjuvant therapy is not considered a systemic regimen
* More than 2 weeks since prior valproic acid
* More than 4 weeks since prior and no concurrent chemotherapy (> 6 weeks for nitrosoureas or mitomycin C) or radiotherapy and recovered

  * Radiotherapy to bone metastasis within the past 2 weeks allowed provided there is active non-bone disease outside the radiation port
* No prior radiotherapy to >= 33% of the bone marrow
* No prior vorinostat or bortezomib
* No concurrent category I medications that are generally accepted to have a risk of causing Torsades de Pointes, including any of the following:

  * Quinidine, procainamide, disopyramide
  * Amiodarone, sotalol, ibutilide, dofetilide
  * Erythromycin, clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients
* No other concurrent investigational agents for the primary malignancy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Attia, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen patients were accrued to this study from June 2009 through July 2010.
Pre-assignment Details: One participant received commercial drug instead of study drug and was deemed a violation. Another participant did not have a post baseline measurement scan and by protocol is not evaluable for the primary endpoint. These patients were excluded from the primary endpoint analysis. Therefore, 14 participants were evaluated for each endpoint.
Period: Overall Study
Arm/Group | Treatment (Vorinostat, Bortezomib)
Started | 16
Completed | 14
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vorinostat, Bortezomib)
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 62 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Tumor Responses
Description: The number of confirmed tumor responses is defined as a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) on two consecutive evaluations at least six weeks apart.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest dimension (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (Vorinostat, Bortezomib)
Number analyzed (Participants) | 14
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival is defined as the time from registration to the time of progression or death, whichever comes first. The distribution and median of progression-free survival times will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vorinostat, Bortezomib)
Number analyzed (Participants) | 14
months | 1.5 [1.3 to 2.9]

3. Secondary Outcome: Overall Survival
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vorinostat, Bortezomib)
Number analyzed (Participants) | 14
months | 16.4 [9.4 to NA] — The upper bound of the 95% confidence interval could not be estimated due to an insufficient number of events.

ADVERSE EVENTS:
Arm/Group | Treatment (Vorinostat, Bortezomib)
Serious Adverse Events (participants affected / at risk) | 6/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat, Bortezomib) (N=16)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat, Bortezomib) (N=16)
Hemoglobin decreased (Blood and lymphatic system disorders) | 12 (35)
Optic nerve edema (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (35)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (35)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 11 (18)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (4)
Fatigue (General disorders) | 15 (48)
Mucosal infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 9 (11)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 13 (33)
Anorexia (Metabolism and nutrition disorders) | 9 (29)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (9)
Peripheral motor neuropathy (Nervous system disorders) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (18)
Syncope (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less